CLINICAL TRIAL: NCT05247255
Title: Quadratus Lumborum (QL) Nerve Block for Patients Undergoing Primary Total Hip Arthroplasty (THA)
Brief Title: Quadratus Lumborum Block for Total Hip Arthroplasty
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Pamela Chia, HS Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-001850
Record Dates: First submitted 2022-01-30; First posted 2022-02-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
Keywords: quadratus lumborum nerve block, analgesia, total hip arthroplasty, postoperative outcomes
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): Quadratus lumborum nerve block with 0.25% ropivacaine
  Interventions: Drug: Active Comparator
- Control Group (Placebo Comparator): Quadratus lumborum nerve block with saline
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Active Comparator — QL block with 0.25% ropivacaine
  Arms: Intervention Group
Drug: Placebo Comparator — QL block with saline
  Arms: Control Group

SUMMARY:
The quadratus lumborum (QL) block is a fascial plane block that has been described to provide analgesia from T7-L3 dermatomes. The investigators aim to evaluate the efficacy of QL blocks in patients undergoing primary total hip arthroplasty (THA).

DETAILED DESCRIPTION:
Investigators will enroll subjects planned for primary THA and allocate them into receiving a QL block with either saline or ropivacaine. Primary outcome will be pain scores over the first 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects undergoing elective primary total hip arthroplasty

Exclusion Criteria:

* patients age < 18,
* documented allergy to local anesthetic
* presence of peripheral neuropathy
* patients with current long term opioid use defined as receiving an opioid on most days in a 90 day period
* patients with a contraindication to spinal and regional anesthesia such as coagulopathy or infection at the site of the regional technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | Up to 48 hrs post op
  Pain scores will be assessed over 48hrs postop using the visual analog score

SECONDARY OUTCOMES:
Opioid usage | Up to 48 hrs post op
  Total morphine-equivalent will be calculated at 0-24hrs and 24-48hrs postop.
Time to first stand | Up to 1 week post surgery
  The period between the end of surgery and the patient's first successful attempt at standing, with or without the assistance of devices (i.e. walker, cane) or staff assistance.
Time to first ambulation | Up to 1 week post surgery
  Time to first ambulation of 50 feet or more, with or without the help of assist devices (i.e. walker, cane) or staff assistance.
Ambulation distance | Up to 1 week post surgery
  This data point will be measured in feet and will be determined by the distance ambulated during the patient's first ambulation attempt after surgery, regardless of the length of ambulation (This distance will be counted regardless of whether the patient reaches the 50 feet requirement to be counted as the "time to first ambulation).
Length of hospital stay | Until discharge from hospital, up to 1 week post surgery
  Number of days in the hospital from postoperative day 0 to discharge
Patient satisfaction | Until day of discharge from the hospital, up to 1 week post surgery
  Patient satisfaction score will be assessed on day of discharge as measured by a 5-point scale with 1 = terrible, 2 = poor, 3 = satisfactory, 4 = good, and 5 = excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Chia, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Santa Monica, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No